CLINICAL TRIAL: NCT01266447
Title: A Phase II Evaluation of ABT-888 (NCI Supplied Agent: ABT-888, NSC #737664), Topotecan (NSC # 609699) and Filgrastim or Pegfilgrastim in the Treatment of Persistent or Recurrent Squamous or Non-squamous Cell Carcinoma of the Cervix
Brief Title: Veliparib, Topotecan Hydrochloride, and Filgrastim or Pegfilgrastim in Treating Patients With Persistent or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02659; NCI-2011-02659 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0127W; CDR0000691281; GOG-0127W (Other: NRG Oncology); GOG-0127W (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma; Recurrent Cervical Carcinoma; Stage III Cervical Cancer; Stage IVA Cervical Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Topotecan; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (veliparib, topotecan hydrochloride, filgrastim) (Experimental): Patients receive veliparib PO twice daily and topotecan hydrochloride IV over 30 minutes once daily on days 1-5. Patients also receive, according to institutional standard, filgrastim SC beginning on day 6, 7, or 8 and continuing until hematopoietic recovery or pegfilgrastim SC on day 6, 7, or 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Biological: Pegfilgrastim; Drug: Topotecan Hydrochloride; Drug: Veliparib

INTERVENTIONS:
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; HSP-130; Neulasta; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Hycamptamine; Hycamtin; SKF S-104864-A; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Veliparib — Given PO
  Other Names: ABT-888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase II clinical trial is studying the how well veliparib, topotecan hydrochloride, and filgrastim or pegfilgrastim work in treating patients with persistent or recurrent cervical cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by blocking them from dividing. Giving veliparib with chemotherapy may kill more tumor cells. Filgrastim or pegfilgrastim may cause the body to make more blood cells and help it recover from the side effects of chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the antitumor activity (objective response rate by RECIST 1.1) of ABT-888 (veliparib) 10 mg administered orally twice a day on days 1 to 5 with topotecan (topotecan hydrochloride) 0.6 mg/m^2 administered IV once daily on days 1 to 5 of each cycle in patients with persistent or recurrent carcinoma of the cervix.

II. To determine the nature and degree of toxicity of ABT-888 and topotecan in patients with persistent or recurrent carcinoma of the cervix.

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free survival and overall survival.

TERTIARY OBJECTIVES:

I. To determine whether evidence of an interaction exists between study treatments and tumor expression of poly(ADP-ribos)ylation of E2 protein, E6/E7 proteins, and p53R2 in relation to progression-free and overall survival or metastasis. (Translational) II. To explore the association between methylation of FanCF and BRCA in pre-treatment tumor samples and pre- and post-treatment biopsy samples and response, progression-free and overall survival of patients, and/or metastasis. (Translational)

OUTLINE:

Patients receive veliparib orally (PO) twice daily and topotecan hydrochloride intravenously (IV) over 30 minutes once daily on days 1-5. Patients also receive, according to institutional standard, filgrastim subcutaneously (SC) beginning on day 6, 7, or 8 and continuing until hematopoietic recovery or pegfilgrastim SC on day 6, 7, or 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples may be collected periodically for translational studies.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have persistent or recurrent squamous cell carcinoma, adenosquamous carcinoma, adenocarcinoma or non-squamous cell carcinoma of the cervix with documented disease progression; histological documentation of the original primary tumor is required via the pathology report
* All patients must have measurable disease as defined by RECIST 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III protocol or Rare Tumor protocol for the same patient population
* Patients must have a GOG performance status of 0, 1, or 2
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Patients should be free of active infection requiring antibiotics
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration; continuation of hormone replacement therapy is permitted
* Any other prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted (non-cytotoxic) therapy and immunologic agents must be discontinued at least three weeks prior to registration; all side effects must have resolved to =< grade 1 or stabilized, prior to enrolling on this study
* Any prior radiation therapy must be completed at least 4 weeks prior to registration
* Patients MUST have had one prior systemic chemotherapeutic regimen for management of advanced, metastatic, or recurrent squamous or non-squamous cell carcinoma of the cervix; chemotherapy administered concurrent with primary radiation is not counted as a systemic chemotherapy regimen (e.g.; weekly cisplatin); adjuvant chemotherapy given following the completion of radiation therapy (or concurrent chemotherapy and radiation therapy) is not counted as a systemic chemotherapy regimen (e.g.; paclitaxel and carboplatin for up to 4 cycles)
* Patients who are registered during the safety lead-in portion of this protocol are required to have prior pelvic radiation
* Patients must have NOT received more than one previous cytotoxic chemotherapy regimen (either with single or combination cytotoxic drug therapy)
* Patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy as part of their one prior systemic chemotherapeutic regimen; patients are allowed to receive, but are not required to receive, biologic/targeted (non-cytotoxic) therapy for management of recurrent or persistent disease
* Patients MUST not be eligible for further curative intent surgical or pelvic radiation treatment for management of recurrent or persistent disease as determined by treating physicians
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* Neuropathy (sensory and motor) less than or equal to grade 1
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have the ability to swallow pills whole

Exclusion Criteria:

* Patients are excluded who have had prior therapy with ABT-888 (veliparib), poly (ADP)-ribose polymerase inhibitors, or topotecan
* Patient with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of cervical cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of cervical cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with seizures or history of seizures are ineligible
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, any CNS metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study, are ineligible; patients with CNS metastases must be stable for > 3 months after treatment and off steroid treatment prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, Principal Investigator — NRG Oncology
Locations (78):
- United States (78):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Decatur Memorial Hospital, Decatur, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - University Medical Center Brackenridge, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - PeaceHealth Medical Group PC, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - D N Greenwald Center, Mukwonago, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 2/7/2011 and closed to accrual on 1/17/2013.
Groups:
- ABT-888, Topotecan and Filgrastim or Pegfilgrastim: ABT-888 10mg administered orally twice a day on days 1 to 5 of each cycle. Topotecan administered at 0.6 mg/m2 intravenously once daily on days 1 to 5 of each cycle. Each cycle of treatment repeats every 21 days until disease progression or adverse effects prohibit further treatment. All patients will receive filgrastim or pegfilgrastim beginning with cycle 1.
Period: Overall Study
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Started | 27
Completed | 27 (Eligible and treated patients)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Complete and Partial Tumor Response as Assessed by RECIST 1.1. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), Complete Response (CR), disappearance of all target and non-target lesions without evidence of new lesion; Partial Response (PR), at least 30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD with no unequivocal progression of non-target lesions and no evidence of new lesion. Complete or partial response requires confirmation at greater than or equal to 4 weeks from initial documentation.
Time Frame: Every other cycle for first 6 months; then every 3 months thereafter until disease progression confirmed; and at any other time if clinically indicted based on symptoms or physical signs suggestive of progressive disease. The average time was 2.3 months
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 27
percentage of participants | 7.4 [2 to 100]

2. Primary Outcome: Number of Patients With Dose-limiting Toxicities (in Safety lead-in)
Description: A dose-limiting toxicity (DLT) is assessed by NCI CTCAE v4, occurring during cycle 1 of therapy.: A dose-limiting toxicity (DLT) is defined as either hematologic or non-hematologic toxicity assessed by NCI CTCAE v4, occurring during cycle 1 of therapy, which cause any of the following: For hematologic toxicity - dose delay of greater than 2 weeks due to failure to recover counts, Treatment related febrile neutropenia, grade 4 neutropenia lasting >7 days, treatment related grade 4 thrombocytopenia or clinically significant bleeding with grade 3 thrombocytopenia. For non-hematologic toxicity; study treatment related grade 3 or 4 non-hematological toxicity (excluding anorexia, constipation, fatigue, hypersensitivity/allergic reaction to one of the study drugs, nausea & vomiting, and grade 3 dehydration), grade 4 nausea and vomiting for >48 hours despite maximum medical management, electrolyte imbalance of > or equal to grade 3 that can be replaced within 48 hours; any drug related death
Time Frame: Up to 21 days
Population: The first 6 eligible and treated patients who completed the 1st cycle of study treatment or had a DLT prior to completing the first cycle of study treatment
Measure: Number; unit: participants
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 6
participants | 1

3. Primary Outcome: Adverse Events (Grade 3 or Higher) During Treatment Period
Description: Number of participants with a maximum grade of 3 or higher during treatment period. Adverse events are graded and categorized using CTCAE v4.0.
Time Frame: During treatment period and up to 30 days after stopping the study treatment.The average of study treatment time was 2.3 months.
Population: Eligible and treated patients - No statistical analysis provided for adverse events (grade 3 or higher) during treatment period.
Measure: Number; unit: Participants
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 27
Participants
  Leukopenia | 6
  Thrombocytopenia | 12
  Neutropenia | 5
  Anemia | 16
  Other Investigations | 4
  Cardiac Disorders | 1
  Gastrointestinal Disorders | 7
  General Disorders & administration site conditions | 5
  Infections and Infestations | 4
  Metabolism and nutrition disorders | 3
  Musculoskeletal and connective tissue disorders | 5
  Neoplasms benign, malignant and unspecified | 1
  Nervous system disorders | 1
  Renal and urinary disorders | 0
  Reproductive system and breast disorders | 2
  Respiratory, thoracic and mediastinal disorders | 4
  Surgical and medical procedures | 1
  Vascular disorders | 3

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the period of time from study entry to time of disease progression, death or date of last contact, whichever occurs first. Progression is defined as at least a 20% increase in the sum of the longest dimensions (LD) of target lesions taking as reference the smallest sum LD recorded since study entry, or unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions, or global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or death due to disease without prior objective documentation of progression.
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first, up to 5 years of follow-up.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 27
months | 2.0 [1.3 to 3.4]

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years of follow-up.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 27
months | 8.2 [5.8 to 10.6]

6. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response is defined as the duration from the time measurement criteria is met for partial or complete response by RECIST 1.1, whichever is first recorded, until the first date the recurrent or progressive disease is objectively documented. Per Response Evaluation Criteria in Solid Tumors (RECIST) criteria Complete Response (CR), disappearance of all target and non-target lesions without evidence of new lesion; Partial Response (PR), at least 30% decrease in the sum of the longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD with no unequivocal progression of non-target lesions and no evidence of new lesion. Complete or partial response requires confirmation at greater than or equal to 4 weeks from initial documentation.
Time Frame: Every other cycle for first 6 months; then every 3 months until disease progression confirmed; and at any other time if clinically indicated based on symptoms or signs suggestive of progressive disease.The average of study treatment time was 2.3 months.
Population: Eligible and Treated Patients with objective response
Measure: Median (Full Range); unit: Months
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Number analyzed (Participants) | 2
Months | 5.3 [4.0 to 6.7]

ADVERSE EVENTS:
Time Frame: During treatment period and up to 30 days after stopping the study treatment. The average of study treatment time was 2.3 months.
Arm/Group | ABT-888, Topotecan and Filgrastim or Pegfilgrastim
Serious Adverse Events (participants affected / at risk) | 16/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-888, Topotecan and Filgrastim or Pegfilgrastim (N=27)
Heart Failure (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Death Nos (General disorders) | 2 (2)
Infections And Infestations - Other (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Respiratory, Thoracic And Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-888, Topotecan and Filgrastim or Pegfilgrastim (N=27)
Anemia (Blood and lymphatic system disorders) | 27
Heart Failure (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Ear And Labyrinth Disorders - Other (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Endocrine Disorders - Other (Endocrine disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 8
Salivary Duct Inflammation (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 7
Rectal Hemorrhage (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 1
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 15
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
General Disorders And Administration Site Conditio (General disorders) | 1
Pain (General disorders) | 7
Malaise (General disorders) | 1
Localized Edema (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 2
Edema Limbs (General disorders) | 2
Fatigue (General disorders) | 22
Fever (General disorders) | 3
Chills (General disorders) | 1
Infections And Infestations - Other (Infections and infestations) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Vaginal Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 5
Lip Infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 4
Weight Loss (Investigations) | 1
Weight Gain (Investigations) | 2
Platelet Count Decreased (Investigations) | 23
Lymphocyte Count Decreased (Investigations) | 4
Inr Increased (Investigations) | 1
Ggt Increased (Investigations) | 1
Creatinine Increased (Investigations) | 3
Neutrophil Count Decreased (Investigations) | 12
Blood Bilirubin Increased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 15
Aspartate Aminotransferase Increased (Investigations) | 2
Alkaline Phosphatase Increased (Investigations) | 8
Alanine Aminotransferase Increased (Investigations) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 9
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Deformity (Musculoskeletal and connective tissue disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal And Connective Tissue Disorder - (Musculoskeletal and connective tissue disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Peripheral Motor Neuropathy (Nervous system disorders) | 2
Memory Impairment (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 3
Dysarthria (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Depressed Level Of Consciousness (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Cystitis Noninfective (Renal and urinary disorders) | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2
Pelvic Pain (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 11
Vascular Disorders - Other (Vascular disorders) | 1
Thromboembolic Event (Vascular disorders) | 4
Lymphedema (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Hot Flashes (Vascular disorders) | 3
Flushing (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less